CLINICAL TRIAL: NCT06003491
Title: A Randomized Controlled Trial for Surgical Treatment of Reducible Atlantoaxial Dislocation
Brief Title: Trial for Surgical Treatment of Reducible Atlantoaxial Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-RCTRAAD
Record Dates: First submitted 2023-07-30; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Atlantoaxial Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular Group (Experimental): Posterior intra-articular distraction and fusion
  Interventions: Device: Intra-articular Cages
- Posterior Group (No Intervention): Posterior direct distraction and fusion

INTERVENTIONS:
Device: Intra-articular Cages — Using reduction using posterior intra-articular distraction and fusion technique with cages.
  Arms: Intra-articular Group

SUMMARY:
The management of reducible atlantoaxial dislocation associated is challenging. Direct posterior distraction technique we proposed in 2010 could achieve satisfactory reduction. In 2020, we modified this technique and proposed a posterior intra-articular distraction technique. The intra-articular distraction technique could theoretically achieve satisfactory reduction and fusion. However, its superiority has not been proven. Therefore, we design a RCT study to compare the reduction rate and fusion rate of different strategies.

ELIGIBILITY:
Inclusion Criteria:

* CT indicated atlantoaxial dislocation Agree with the operation plan Agree to be followed up

Exclusion Criteria:

* The pathology is traumatic or RA Underwent operations in occipital-cervical region before With mortal diseases Without ability to sign papers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Fusion Rates | 12 months
  Atlantoaixal fusion rates

SECONDARY OUTCOMES:
Japanese Orthopaedic Association Scores | 12 months
  0-17 Scores
Visual Analogue Scale | 12 months
  0-10 Scores
Neck Disability Index | 12 months
  0-5 Scores

REFERENCES:
- [Background] Chen Z, Duan W, Chou D, Guan J, Liu Z, Jian Q, Zhang B, Bo X, Jian F. A Safe and Effective Posterior Intra-Articular Distraction Technique to Treat Congenital Atlantoaxial Dislocation Associated With Basilar Invagination: Case Series and Technical Nuances. Oper Neurosurg. 2021 Mar 15;20(4):334-342. doi: 10.1093/ons/opaa391. PMID 33372978